CLINICAL TRIAL: NCT01794689
Title: Mechanisms of Sleep Disruption Hyperalgesia
Acronym: ESP2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: NA_00071465; 1R01DA032922-01 (NIH)
Record Dates: First submitted 2013-02-15; First posted 2013-02-20 (Estimated); Results first posted 2019-02-22 (Actual); Last update posted 2019-08-02 (Actual); Status verified 2019-08

CONDITIONS: Sleep Deprivation; Pain
MeSH Terms: conditions — Sleep Deprivation; Pain | interventions — Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (4):
- Morphine US then Morphine FA (Experimental): Participants randomized to receive Morphine and the Uninterrupted Sleep (US) condition first. After a polysomnography (PSG) screening night, participants were randomized to receive two consecutive nights of uninterrupted sleep (US). With a minimum of a two week washout period, participants then completed the opposing sleep condition of two nights of forced awakenings (FA). They will receive the Morphine injection (0.08mg/kg) via IV bolus over 30 seconds during each experimental quantitative sensory testing session that occurs after the US and FA sleep conditions are completed.
  Interventions: Drug: Morphine; Behavioral: Forced Awakenings; Behavioral: Uninterrupted Sleep
- Placebo US then Placebo FA (Placebo Comparator): Participants randomized to receive the saline placebo and the Uninterrupted Sleep (US) condition first. After a polysomnography (PSG) screening night, participants were randomized to receive two consecutive nights of uninterrupted sleep (US). With a minimum of a two week washout period, participants then completed the opposing sleep condition of two nights of forced awakenings (FA). They will receive the injection via IV bolus over 30 seconds during each experimental quantitative sensory testing session that occurs after the US and FA sleep conditions are completed.
  Interventions: Drug: Saline Placebo; Behavioral: Forced Awakenings; Behavioral: Uninterrupted Sleep
- Morphine FA then Morphine US (Experimental): Participants randomized to receive Morphine and the Forced Awakenings (FA) condition first. After a polysomnography (PSG) screening night, participants were randomized to receive two consecutive nights of forced awakenings (FA). With a minimum of a two week washout period, participants then completed the opposing sleep condition of two nights of uninterrupted sleep (US). They will receive the Morphine injection (0.08mg/kg) via IV bolus over 30 seconds during each experimental quantitative sensory testing session that occurs after the FA and US sleep conditions are completed.
  Interventions: Drug: Morphine; Behavioral: Forced Awakenings; Behavioral: Uninterrupted Sleep
- Placebo FA then Placebo US (Placebo Comparator): Participants randomized to receive the saline placebo and the Forced Awakenings (FA) condition first. After a polysomnography (PSG) screening night, participants were randomized to receive two consecutive nights of forced awakenings (FA). With a minimum of a two week washout period, participants then completed the opposing sleep condition of two nights of uninterrupted sleep (US). They will receive the injection via IV bolus over 30 seconds during each experimental quantitative sensory testing session that occurs after the FA and US sleep conditions are completed.
  Interventions: Drug: Saline Placebo; Behavioral: Forced Awakenings; Behavioral: Uninterrupted Sleep

INTERVENTIONS:
Drug: Morphine — 0.08mg/kg will be administered to participants randomly assigned to receive the drug via IV bolus during each quantitative sensory testing session (after one night of uninterrupted sleep and after 2 nights of forced awakenings).
  Arms: Morphine FA then Morphine US; Morphine US then Morphine FA
Drug: Saline Placebo — Saline Placebo will administered to participants randomly assigned to receive the placebo via IV bolus during each quantitative sensory testing session (after one night of uninterrupted sleep and after 2 nights of forced awakenings).
  Arms: Placebo FA then Placebo US; Placebo US then Placebo FA
Behavioral: Forced Awakenings — Participants will be awakened each hour during an 8 hour sleep opportunity period. One of the awakenings is for 60 minutes and randomly determined. The other 7 awakenings are for 20 minutes each, and are randomly scheduled to occur in either the first second or third tertile of each hour. The maximum total sleep time a participant will receive is 280 minutes.
Behavioral: Uninterrupted Sleep — Participants will receive an 8 hour period of undisturbed sleep

SUMMARY:
Twenty percent of Americans suffer from chronic pain. Sleep disturbance is similarly prevalent and among the most common and disabling neurobehavioral problems associated with chronic pain. This research is designed to evaluate the effects of disrupted sleep patterns on mood, inflammation, the perception of pain, and pain relief. This study will help researchers understand the relationship between sleep and pain, and how sleep disturbance might influence chronic pain conditions.

DETAILED DESCRIPTION:
This research is being conducted in order to evaluate the effects of disrupted sleep patterns on mood, inflammation, the perception of pain, and pain relief. This study will help researchers understand the relationship between sleep and pain, and how sleep disturbance might influence chronic pain conditions. Healthy participants will undergo baseline sleep and sleep disruption conditions. Following undisturbed sleep and sleep disruption conditions, sensitivity to pain and analgesic response (via morphine or placebo administration) will be assessed using a heat-capsaicin pain model.

This study will be conducted in 2 major parts-3 screening visits (2 outpatient and 1 inpatient) and 2 experimental inpatient visits. Part 1 of the study will involve a 1-week screening period. This will involve two separate screening visits lasting about 2 hours each. At Screening Visit 1, participants will complete questionnaires, an interview, and undergo toxicology screening. At Screening Visit 2, participants will complete questionnaires, undergo a physical exam, and be familiarized with pain testing procedures. At Screening Visit 3, participants will undergo an inpatient sleep study.

Part 2 will involve two different inpatient admissions. The two admissions will be separated by at least two weeks. During each of the admissions, participants' sleep will be studied at night. The first admission will begin immediately following the overnight sleep study in Screening Visit 3. One of the admissions will be for one night and the other admission will be for three nights. For the one night admission, participants will sleep undisturbed for an 8-hour period. For the three night admission, participants will undergo sleep disruption for two nights in a row. On the third night, participants will be allowed to sleep undisturbed for 8 hours for recovery.

During both inpatient admissions, pain testing procedures will be completed that will last approximately 5 hours during the day. During testing, small amounts of blood will be drawn for analysis. Participants will be randomly assigned to two groups. Group A will be given a standard dose of morphine during pain testing. Group B will be given a placebo during pain testing.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Age 18-48
* Meets Research Diagnostic Criteria for Normal Sleepers
* Stable sleep phase within 21:00 and 08:00
* Total sleep time between 6.5 and 8.5 hours per night
* Sleep efficiency ≥85%
* Epworth Sleepiness Scale Score <10
* Non-smoker/non-nicotine users
* Low Caffeine Users (≤2 cups per day)

Exclusion Criteria:

* Body Mass Index ≥35
* Lifetime history of chronic pain (>6 months)
* Acute pain
* Significant medical or psychiatric morbidity within 6 months
* Lifetime history of bipolar disorder, psychotic disorder, serious recurrent major depression, serious post-traumatic stress disorder, or seizure disorder
* Respiratory, hepatic, renal, or cardiac conditions that would contraindicate opioid use
* Lifetime history of alcohol or substance abuse or dependence
* Lifetime history of opioid use >36 doses or >7 days of consecutive use
* Prior adverse reaction to general anesthetics, opioids, or capsaicin
* Clinically significant abnormal complete blood count or comprehensive metabolic profile
* Positive toxicology screen for opioids or recreational drugs
* Pregnant or lactating women
* Significant pre-admission psychological distress (T-scores >64 on the Brief Symptom Inventory Global Scales)
* Significant lifetime history of serious head injury that is determined to influence pain processing or sleep systems

Ages: 18 Years to 48 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2019-03-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Smith, Ph.D, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University Bayview Medical Center, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Irwin MR, Olmstead R, Bjurstrom MF, Finan PH, Smith MT. Sleep disruption and activation of cellular inflammation mediate heightened pain sensitivity: a randomized clinical trial. Pain. 2023 May 1;164(5):1128-1137. doi: 10.1097/j.pain.0000000000002811. Epub 2022 Oct 27. PMID 36314570

RESULTS

PARTICIPANT FLOW:
Recruitment Details: During screening for the study we evaluated whether participants were generally healthy, pain free, and good sleepers. We screened 255 to obtain 100 participants who met criteria and were randomized to the experimental portion of the study. The experimental phase occurred at an inpatient clinical research unit.
Period: Intervention 1 (2 Nights)
Arm/Group | Morphine US Then Morphine FA | Morphine FA Then Morphine US | Placebo US Then Placebo FA | Placebo FA Then Placebo US
Started | 25 | 29 | 24 | 22
Completed | 20 | 27 | 21 | 18
Not Completed | 5 | 2 | 3 | 4
Not completed — Withdrawal by Subject | 3 | 0 | 2 | 4
Not completed — Protocol Violation | 1 | 0 | 1 | 0
Not completed — Physician Decision | 1 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0
Period: Washout (2 Weeks)
Arm/Group | Morphine US Then Morphine FA | Morphine FA Then Morphine US | Placebo US Then Placebo FA | Placebo FA Then Placebo US
Started | 20 | 27 | 21 | 18
Completed | 20 | 27 | 21 | 18
Not Completed | 0 | 0 | 0 | 0
Period: Intervention 2 (2 Nights)
Arm/Group | Morphine US Then Morphine FA | Morphine FA Then Morphine US | Placebo US Then Placebo FA | Placebo FA Then Placebo US
Started | 20 | 27 | 21 | 18
Completed | 20 | 27 | 21 | 18
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Morphine US Then Morphine FA | Morphine FA Then Morphine US | Placebo US Then Placebo FA | Placebo FA Then Placebo US | Total
Number analyzed (Participants) | 25 | 29 | 24 | 22 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.1348 (5.97835) | 29.6819 (7.54226) | 27.3609 (5.22747) | 27.7272 (8.18124) | 28.0581 (6.81392)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 15 | 12 | 17 | 58
  Male | 11 | 14 | 12 | 5 | 42
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 3 | 6 | 1 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 10 | 10 | 6 | 11 | 37
  White | 10 | 14 | 11 | 10 | 45
  More than one race | 3 | 0 | 0 | 0 | 3
  Unknown or Not Reported | 1 | 2 | 1 | 0 | 4
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 26.1490 (4.16713) | 25.2645 (3.95007) | 25.8440 (3.63156) | 25.7134 (4.17552) | 25.7235 (3.93648)

OUTCOME MEASURES:

1. Primary Outcome: Spinal Sensitization as Assessed by Area of Secondary Hyperalgesia (2HA) After Two Nights of Uninterrupted Sleep and Two Nights of 8 Forced Awakenings
Description: The area of secondary hyperalgesia (2HA) to mechanical stimulation was quantified by stimulating along eight linear paths near the capsaicin treated site using a 15 gram nonpainful von Frey filament. Stimulation occurred until the participant reported a change in sensation from which a border was marked on the skin. The degree of 2HA was assessed by measuring the total surface area (mm^2) of the marked borders. Data were collapsed by group to analyze the effects of FA vs US, irrespective of randomization group. Our Primary Secondary Hyperalgesia outcome was measured prior to injection of either morphine or placebo.
Time Frame: Next day during quantitative sensory testing after 2 nights of forced awakenings or uninterrupted sleep
Measure: Mean (Standard Deviation); unit: mm^2
Groups:
- Morphine US: Participants that received morphine with Uninterrupted sleep (US).
- Morphine FA: Participants that received morphine with forced awakenings (FA).
- Placebo US: Participants that received placebo with Uninterrupted sleep (US).
- Placebo FA: Participants that received placebo with forced awakenings (FA).
Arm/Group | Morphine US | Morphine FA | Placebo US | Placebo FA
Number analyzed (Participants) | 47 | 47 | 39 | 39
mm^2 | 1276.25 (1096.761) | 1582.67 (1590.784) | 1302.93 (1301.457) | 1447.9 (1322.52)

2. Secondary Outcome: Opioid Analgesia as Assessed by Analgesia Index (Seconds)
Description: After 2 nights of forced awakenings and after two nights of uninterrupted sleep, opioid analgesia will be assessed by an analgesia index. The analgesia index is calculated using withdrawal latency during cold pressor testing (lasting maximum of 300 seconds). Cold Pressor Testing is done before and after morphine or placebo injection. The difference in withdrawal time before and after morphine or placebo injection is the analgesia index with a minimum score of -300 seconds and maximum score of 300 seconds. These data were log transformed. Mean analgesia index was then calculated for each group. Higher means represent greater analgesia.
Time Frame: Next day after 2 nights of forced awakenings or uninterrupted sleep
Population: Each participant had to do four visits and two testing sessions to be termed complete. The data needed for analysis for this outcome measure was obtained from some participants but not all who completed or couldn't complete the entire study. This explains the differences in the number of units analyzed.
Measure: Mean (Standard Deviation); unit: seconds (log transformed)
Units Other Than Participants: cold pressor test
Arm/Group | Morphine US | Morphine FA | Placebo US | Placebo FA
Number analyzed (Participants) | 47 | 47 | 39 | 39
Number analyzed (cold pressor test) | 48 | 45 | 42 | 39
seconds (log transformed) | 0.315 (0.540) | 0.156 (0.712) | -0.124 (0.346) | -0.006 (0.263)

3. Secondary Outcome: Mean Change in Percentage of Peripheral Blood Mononuclear Cells Expressing Interleukin-6 After LPS Stimulation
Description: After 2 nights of forced awakenings, and two nights of uninterrupted sleep, blood is drawn (approximately every 60 minutes) during quantitative sensory testing; 4 hours pre-morphine/placebo administration and 2 hours post-morphine/placebo administration to examine markers of inflammation. Two blood samples for each participant are analyzed at 7 separate time points. The marker of inflammation assessed is the number of peripheral blood mononuclear cells expressing Interleukin-6 (IL-6), and the outcome measure represents the mean change in IL-6 levels pre and post stimulation with lipopolysaccharide (LPS). Cellular IL-6 expression was was quantified via flow cytometry.
Time Frame: Next day after 2 nights of forced awakenings or uninterrupted sleep, every 60 minutes up to 7 hours
Population: For some participants we could not collect blood samples for all time points and testing sessions. This explains the differences in the numbers of samples analyzed at various timepoints.
Measure: Mean (Standard Deviation); unit: percentage of IL-6 expression
Units Other Than Participants: blood samples
Arm/Group | Morphine US | Morphine FA | Placebo US | Placebo FA
Number analyzed (Participants) | 47 | 47 | 39 | 39
Number analyzed (blood samples) | 265 | 256 | 225 | 213
percentage of IL-6 expression
  Timepoint 1: number analyzed (blood samples) | 38 | 38 | 31 | 32
  Timepoint 1 | 41.98 (21.18) | 51.82 (21.13) | 42.91 (19.53) | 43.32 (19.04)
  Timepoint 2: number analyzed (blood samples) | 38 | 37 | 32 | 32
  Timepoint 2 | 45.44 (22.95) | 51.84 (20.34) | 42.93 (21.81) | 43.79 (18.01)
  Timepoint 3: number analyzed (blood samples) | 38 | 37 | 34 | 32
  Timepoint 3 | 45.99 (19.12) | 48.99 (18.96) | 40.76 (20.1) | 41.65 (21.87)
  Timepoint 4: number analyzed (blood samples) | 38 | 38 | 34 | 32
  Timepoint 4 | 43.96 (18.2) | 46.94 (17.81) | 39.06 (20.48) | 41.34 (21.36)
  Timepoint 5: number analyzed (blood samples) | 38 | 35 | 33 | 31
  Timepoint 5 | 38.67 (17.93) | 43.45 (18.3) | 38.71 (19.11) | 34.63 (20.74)
  Timepoint 6: number analyzed (blood samples) | 38 | 36 | 31 | 27
  Timepoint 6 | 36.83 (19.39) | 39.15 (21.23) | 35.64 (18.58) | 36.28 (19.38)
  Timepoint 7: number analyzed (blood samples) | 37 | 35 | 29 | 27
  Timepoint 7 | 36.47 (18.9) | 39.92 (19.6) | 35.49 (17.03) | 35.25 (19.35)

4. Other Pre Specified Outcome: Total Sleep Time
Description: The degree of sleep deprivation will be assessed by total sleep time (TST) in minutes during the uninterrupted sleep condition compared to the forced awakenings conditions.
Time Frame: Next day during quantitative sensory testing after 2 nights of forced awakenings or uninterrupted sleep.
Population: Each participant had to do four visits to be termed complete. The data needed for analysis for this outcome measure was obtained from some participants but not all who completed or couldn't complete the entire study. This explains the differences in the numbers analyzed for each total sleep time.
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- Morphine US: Participants randomized to receive Morphine and the Uninterrupted Sleep (US) condition first. After a polysomnography (PSG) screening night, participants were randomized to receive two consecutive nights of uninterrupted sleep (US). With a minimum of a two week washout period, participants then completed the opposing sleep condition of two nights of forced awakenings (FA). They will receive the Morphine injection (0.08mg/kg) via IV bolus over 30 seconds during each experimental quantitative sensory testing session that occurs after the US and FA sleep conditions are completed.
- Morphine FA: Participants randomized to receive Morphine and the Forced Awakenings (FA) condition first. After a polysomnography (PSG) screening night, participants were randomized to receive two consecutive nights of forced awakenings (FA). With a minimum of a two week washout period, participants then completed the opposing sleep condition of two nights of uninterrupted sleep (US). They will receive the Morphine injection (0.08mg/kg) via IV bolus over 30 seconds during each experimental quantitative sensory testing session that occurs after the FA and US sleep conditions are completed.
- Placebo US: Participants randomized to receive the saline placebo and the Uninterrupted Sleep (US) condition first. After a polysomnography (PSG) screening night, participants were randomized to receive two consecutive nights of uninterrupted sleep (US). With a minimum of a two week washout period, participants then completed the opposing sleep condition of two nights of forced awakenings (FA). They will receive the injection via IV bolus over 30 seconds during each experimental quantitative sensory testing session that occurs after the US and FA sleep conditions are completed.
- Placebo FA: Participants randomized to receive the saline placebo and the Forced Awakenings (FA) condition first. After a polysomnography (PSG) screening night, participants were randomized to receive two consecutive nights of forced awakenings (FA). With a minimum of a two week washout period, participants then completed the opposing sleep condition of two nights of uninterrupted sleep (US). They will receive the injection via IV bolus over 30 seconds during each experimental quantitative sensory testing session that occurs after the FA and US sleep conditions are completed.
Arm/Group | Morphine US | Morphine FA | Placebo US | Placebo FA
Number analyzed (Participants) | 25 | 29 | 24 | 22
minutes
  TST: Uninterrupted Sleep-Night 1: number analyzed (Participants) | 22 | 25 | 24 | 15
  TST: Uninterrupted Sleep-Night 1 | 442.8909 (23.06461) | 425.0280 (52.40921) | 443.2375 (38.99631) | 435.1467 (29.12669)
  TST: Uninterrupted Sleep-Night 2: number analyzed (Participants) | 22 | 24 | 24 | 15
  TST: Uninterrupted Sleep-Night 2 | 435.2045 (41.16120) | 420.1375 (71.39364) | 439.0417 (47.06713) | 441.1400 (35.93814)
  TST: Forced Awakenings-Night 1: number analyzed (Participants) | 18 | 26 | 22 | 20
  TST: Forced Awakenings-Night 1 | 217.4556 (46.00094) | 225.4192 (38.47452) | 235.1727 (50.91526) | 252.0950 (32.70550)
  TST: Forced Awakenings-Night 2: number analyzed (Participants) | 18 | 24 | 21 | 17
  TST: Forced Awakenings-Night 2 | 270.3333 (35.23125) | 258.1083 (29.47026) | 267.7714 (16.90080) | 261.9941 (32.01372)

ADVERSE EVENTS:
Time Frame: Participants were enrolled and actively participating in the study across a time frame of four years and 7.5 months. With no scheduling difficulties each participant remained in the study for 5-6 weeks.
Arm/Group | Morphine US | Morphine FA | Placebo US | Placebo FA
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/49 | 0/42 | 0/43
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/49 | 0/42 | 0/43
Other Adverse Events (participants affected / at risk) | 8/52 | 7/49 | 1/42 | 2/43
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Morphine US (N=52) | Morphine FA (N=49) | Placebo US (N=42) | Placebo FA (N=43)
Hypotension (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 6 (8) | 5 (8) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 4 (5) | 5 (9) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 3 (3) | 2 (4) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Stomach Pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Laceration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Claustrophobia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Participants were mostly young adults, were generally healthy, pain free and good sleepers. Strict inclusion/exclusion criteria and high participant burden (laboratory pain testing, overnight sleep studies) impacted sample size and study completion.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-30): https://cdn.clinicaltrials.gov/large-docs/89/NCT01794689/Prot_SAP_000.pdf